CLINICAL TRIAL: NCT06627855
Title: Investigation of the Effectiveness of Manual Therapy Based on Fascial Distortion Model in Individuals With Temporomandibular Disorder: A Randomized Sham-controlled Trial
Brief Title: Effectiveness of the Fascial Distortion Model in Temporomandibular Disorders: A Randomized Sham-controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Harun Gençosmanoğlu, Lecturer, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/1627
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Disorders (TMD); Manual Therapy; Fascial Distortion
Keywords: manual therapy; fascial distortion model; temporomandibular disorders; head posture
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Therapy based Fascial Distortion Model (Active Comparator): It will conducted for forty-five minutes once a week in a clinical setting for 4 weeks.
  Interventions: Procedure: Fascial Distortion Model
- Control (Sham Comparator): Sham application will conducted for forty-five minutes once a week in a clinical setting for 4 weeks.
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Fascial Distortion Model — The following techniques were used on the cranial and cervical areas during therapy: Trigger band technique, herniated trigger point technique, continuum technique, folding technique, cylinder technique, and tectonic technique.
  Other Names: Typaldos Manual Therapy
  Arms: Manual Therapy based Fascial Distortion Model
Procedure: Sham treatment — The techniques in the therapy will be applied by imitating the techniques in the therapy for the fascial distortions determined according to the Manual Therapy Based on the Fascial Distortion Model.
  Arms: Control

SUMMARY:
The aim of the study was to investigate the effectiveness of Manual Therapy Based on the Fascial Distortion Model in individuals with temporomandibular disorders compared to sham control. Individuals diagnosed with temporomandibular disorder will be randomly assigned to groups as Group 1 (Manual Therapy Based on Fascial Distortion Model) and Group 2 (Sham Control). Head posture, cervical and temporomandibular joint range of motion, cervical muscle performance, pain intensity, pressure pain thresholds, temporomandibular disorder severity, disability, dysfunction, health-related quality of life, kinesiophobia, and central sensitization will be assessed.

DETAILED DESCRIPTION:
Interventions are needed to address head posture, cervical and temporomandibular joint range of motion, cervical muscle performance, pain intensity, pressure pain thresholds, temporomandibular disorder severity, disability, dysfunction, health-related quality of life, kinesiophobia, and central sensitization in individuals with temporomandibular disorder (TMD). This study aims to examine the effectiveness of Manual Therapy Based on the Fascial Distortion Model in individuals with TMDs compared to sham control over a 4-week period. Individuals with TMD will be randomized into Group 1 (Fascial Distortion Model-based Manual Therapy) or Group 2 (Sham Control). Interventions will be conducted once a week in a clinical setting. Head posture will be measured by lateral photogrammetry, cervical range of motion will be measured by an inclinometer, temporomandibular range of motion will be measured by a vernier caliper, cervical muscle performance will be measured by Cervical Spine Functional Strength Test, and pressure pain threshold will be measured by an algometer. Pain intensity will be assessed using the Graded Chronic Pain Scale (Revised) and the Short-Form McGill Pain Questionnaire. TMD severity will be assessed using the Fonseca Anamnestic Index. Mandibular Function Impairment Questionnaire will be used to assess dysfunction. Disability will be evaluated using the Craniofacial Pain and Disability Inventory. Health-related quality of life will be assessed using Short Form-36. Kinesiophobia will be assessed with the Tampa Kinesiophobia Scale; central sensitization will be assessed with the Central Sensitisation Inventory.

All outcomes will be measured at baseline and end of the study, while pain intensity and pressure pain thresholds will also undergo intermediate assessments (2nd and 3rd week).

ELIGIBILITY:
Inclusion Criteria:

* Having temporomandibular joint complaints and being diagnosed with temporomandibular disorder according to the Diagnostic Criteria for Temporomandibular Disorders Axis I
* Understand and be willing to answer assessment questions
* A temporomandibular joint complaint for the last three months
* Pain in the jaw, face or neck

Exclusion Criteria:

* Has a systemic disease (neurological, rheumatologic, oncologic, etc.) that may affect the temporomandibular joint, cervical spine and/or assessment
* Any history of trauma that may have affected the cranio-cervico-facial region
* Having undergone any surgical intervention in the cranio-cervico-facial region within the last six months
* Receiving surgical treatment, medical treatment, splint therapy or physiotherapy for temporomandibular disorder in the last month
* Radiotherapy in the head and neck region
* Pregnancy or breastfeeding
* Exercise therapy for craniocervical posture for the last month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Head posture | From enrollment to the end of treatment at 4th week
  Lateral photogrammetry according to Eye-Tragus-Horizontal Angle, Pogonion-Tragus-C7 Angle, Tragus-C7-Horizontal Angle, Tragus-C7-Shoulder Angle, and Shoulder-C7-Horizontal Angle.
Cervical range of motions | From enrollment to the end of treatment at 4th week
  Inclinometric measurements based on flexion, extension, lateral flexions, and rotations.
Temporomandibular range of motions | From enrollment to the end of treatment at 4th week
  Digital vernier caliper measurements based on maximum pain-free mouth opening, maximum possible mouth opening, maximum possible assisted mouth opening, laterotrusions, and protrusion.
Cervical muscle performance | From enrollment to the end of treatment at 4th week
  The Functional Strength Testing of the Cervical Spine was used to evaluate the cervical muscle performance. This is a test that functionally evaluates cervical muscle strength. Results of this test are assessed as functional, functionally fair, functionally poor, and nonfunctional. Six-to-eight repetitions for the flexion test and 20-25 s holding time for the other tests indicate that the test result is functional. Three-to-five repetitions for the flexion test and 10-19 s holding time for the other tests indicate that the test result is functionally fair. One-to-two repetitions for the flexion test and 1-9 s holding time for the other tests indicate that the test result is functionally poor. Zero repetition for the flexion test and 0 s holding time for the other tests indicate that the test result is nonfunctional. Each test was terminated at onset of pain, and the relevant value was recorded.
Pressure pain threshold | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Algometer. Tempormandibular joint, masseter, temporalis anterior, suboccipital muscle, trapezius, lateral epicondyle for both side.
Pain intensity in the last week | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Short-Form McGill Pain Questionnaire. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Chronic pain intensity | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Graded Chronic Pain Scale (Revised). Scoring: Grade 1=mild, Grade 2=bothersome, Grade 3=high impact chronic pain. Higher scores mean a worse outcome.
Temporomandibular disorders severity | From enrollment to the end of treatment at 4th week
  Fonseca Anamnestic Index. Minimum and maximum values are 0 and 10 points, respectively. Higher scores mean a worse outcome.
Dysfunction | From enrollment to the end of treatment at 4th week
  Mandibular Function Impairment Questionnaire. Minimum and maximum values are 0 and 4 points, respectively. Higher scores mean a worse outcome.
Disability | From enrollment to the end of treatment at 4th week
  Craniofacial Pain and Disability Inventory. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Health-related quality of life | From enrollment to the end of treatment at 4th week
  Short Form-36. Its subdomains are physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
Kinesiophobia | From enrollment to the end of treatment at 4th week
  Tampa Kinesiophobia Scale for Temporomandibular Disorders. Minimum and maximum values are 1 and 4 points, respectively. Higher scores mean a worse outcome.
Central sensitization | From enrollment to the end of treatment at 4th week
  Central Sensitisation Inventory. Minimum and maximum values are 0 and 4 points, respectively. Higher scores mean a worse outcome.
Present pain intensity | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Visual Analog Scale. Minimum and maximum values are 0 and 10 cm, respectively. Higher scores mean a worse outcome.
Present pain intensity (ordinal) | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Present pain intensity scale of McGill Pain Questionnaire. Minimum and maximum values are 0 and 5 points, respectively. Higher scores mean a worse outcome.
Pain intensity in the last week (ordinal) | From enrollment to the end of treatment at 1st week, 2nd week, 3rd week, and 4th week.
  Numeric Pain Rating Scale. Minimum and maximum values are 0 and 10 points, respectively. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Harun Gençosmanoğlu, PT, MSc, Principal Investigator — Karabük University
Locations (1):
- Karabük University, Merkez, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No